CLINICAL TRIAL: NCT04398433
Title: An Open-label Multi-center Study of INO-3107 With Electroporation (EP) in Subjects With HPV-6- and/or HPV-11-associated Recurrent Respiratory Papillomatosis (RRP)
Brief Title: INO-3107 With Electroporation (EP) in Participants With HPV-6- and/or HPV-11-Associated Recurrent Respiratory Papillomatosis (RRP)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Inovio Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRP-001
Record Dates: First submitted 2020-05-14; First posted 2020-05-21 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Respiratory Papillomatosis
Keywords: Human papilloma virus (HPV)
MeSH Terms: conditions — Recurrent respiratory papillomatosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- INO-3107 (Experimental): Participants will be administered one INO-3107 intramuscular (IM) injection followed by electroporation (EP) using CELLECTRA™ 2000 at Day 0, Week 3, Week 6, and Week 9.
  Interventions: Drug: INO-3107; Device: CELLECTRA™ 2000

INTERVENTIONS:
Drug: INO-3107 — INO-3107 administered by IM injection followed by EP using CELLECTRA™ 2000 device at Day 0, Week 3, 6, and 9.
Device: CELLECTRA™ 2000 — CELLECTRA™ 2000 device used for EP following IM delivery of INO-3107.

SUMMARY:
This is a Phase 1/2 open-label, multicenter trial to evaluate the safety, tolerability, immunogenicity, and efficacy of INO-3107 in subjects with HPV-6 and/or HPV-11-associated recurrent respiratory papillomatosis (RRP). The trial population will include participants who have been diagnosed with either Juvenile-Onset RRP (J-O RRP) as defined by age at first diagnosis <12 years or with Adult- Onset RRP (A-O RRP) as defined by age at first diagnosis ≥12 years. A safety run-in will be performed with up to six participants with a one week waiting period between each enrolled participant.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically-documented HPV-6- or HPV-11-positive respiratory papilloma or documentation of low-risk positive HPV using a Sponsor approved HPV-6/11 type-specific assay
* Requirement for frequent RRP intervention to remove or resect respiratory papilloma, as defined as at least two RRP surgical (including laser) interventions in the year prior to and including Day 0
* Must be an appropriate candidate for upcoming surgical intervention as per Investigator judgment and RRP Staging Assessment score
* Adequate bone marrow, hepatic, and renal function
* Participants must meet one of the below requirements:

  * Be of non-child bearing potential (≥12 months of non-therapy-induced amenorrhea, confirmed by follicle-stimulating hormone [FSH], if not on hormone replacement)
  * Be surgically sterile (vasectomy in males or absence of ovaries and/or uterus in females)
  * Agree to use one highly effective or combined contraceptive methods that result in a failure rate of <1% per year during the treatment period and at least through week 12 after last dose
  * Agree to abstinence from penile-vaginal intercourse, when this is the participant's preferred and usual lifestyle

Key Exclusion Criteria:

* Recipient of therapy directed towards RRP disease (other than surgery or ablation) including but not limited to anti-virals (including cidofovir), radiation, chemotherapy, anti-angiogenic therapy (including bevacizumab), prophylactic HPV vaccination (including Gardasil) as therapeutic intervention, or therapy with an experimental agent within 3 months prior to Day 0
* Ongoing or recent (within 1 year) evidence of autoimmune disease that required treatment with systemic immunosuppressive treatments, with the exception of: vitiligo, childhood asthma that has resolved, type 1 diabetes, residual hypothyroidism that requires only hormone replacement, or psoriasis that does not require systemic treatment
* Diagnosis of immunodeficiency or treatment with systemic immunosuppressive therapy within 28 days prior to the first dose of trial treatment, including systemic corticosteroids
* High risk of bleeding or require the use of anticoagulants for management of a known bleeding diathesis
* Recipient of any live virus vaccine within 4 weeks prior to the first dose of trial treatment or any non-live vaccine within two weeks prior to the first dose of trial treatment
* History of clinically significant, medically unstable disease which, in the judgment of the Investigator, would jeopardize the safety of the participant, interfere with trial assessment or evaluation, or otherwise impact the validity of the trial results
* Fewer than two acceptable sites are available for IM injection considering the deltoid and anterolateral quadriceps muscles. Study treatment should not be given within 2 centimeters (cm) of a tattoo, keloid or hypertrophic scar. If there is implanted metal, implanted device, within the same limb the use of the deltoid muscle on the same side of the body is excluded
* Prisoners or participants who are compulsory detained (involuntary incarceration) for treatment of either a psychiatric or physical (i.e. infectious disease) illness
* Any medical or psychological or non-medical condition that might interfere with the participation or safety of the participant, as determined by the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) and Serious Adverse Events (SAEs) | Screening up to Week 52 (up to approximately 1 year)
  An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. An AE can include any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product. A serious adverse event (SAE) is any untoward medical occurrence that at any dose: 1. Results in death. 2. A life-threatening event; however, this does not include an event that, had it occurred in a more severe form, might have caused death. 3. Requires inpatient hospitalization or prolongation of existing hospitalization. 4. Results in persistent or significant disability/incapacity. 5. Results in a congenital anomaly/birth.

SECONDARY OUTCOMES:
The Number of RRP Surgical Interventions in the 52 Weeks Post Day 0 Compared to the Number of RRP Surgical Interventions in the Year Prior to Day 0 Dosing | Screening up to Week 52 (up to approximately 1 year)
Change in RRP Staging Assessment Scores Over Time | Screening, Day 0, Weeks 6, 11, 26, 52 (up to approximately 1 year)
  An RRP Staging Assessment score will be determined using a modified Derkay staging tool. It includes both a subjective functional assessment of clinical parameters and an anatomic assessment of disease distribution. The anatomic score can then be used in combination with the functional score to measure an individual patient's clinical course and response to the therapy over time.
Change from Baseline in Interferon-gamma Enzyme-Linked Immunosorbent Spot (IFN-γ ELISpot) Response Magnitude for IFN-γ Secreting Cells in Peripheral Blood Mononuclear Cells (PBMCs) | Baseline, Weeks 6, 9, 11, 26, 52
Change from Baseline in Flow Cytometry Response Magnitude for T-cell Phenotype and Lytic Potential in PBMCs | Baseline, Weeks 6, 9, 11, 26, 52
Change from Baseline in Resected Tumor Tissue Response Magnitude for Pro-inflammatory and Immunosuppressive Elements | Baseline and at subsequent tissue resections, up to Week 52 (up to approximately 1 year)
Change from Baseline in MicroRNA (miRNA) Expression Related to Reduced Frequency of RRP Surgical Intervention | Baseline and Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Skolnik, MD, Study Director — Inovio Pharmaceuticals
Locations (11):
- United States (11):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - University of California at Davis, Sacramento, California
  - Winship at Emory University Hospital Midtown, Atlanta, Georgia
  - Johns Hopkins University School of Medicine, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - NYU Langone Voice Center, New York, New York
  - UNC School of Medicine, Chapel Hill, North Carolina
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data dictionaries and all collected IPD will be stripped of identifiers and may be made available upon request.
Supporting Information: Study Protocol, ICF
Time Frame: Anonymous IPD may be shared following or during the publication of summary data. Archival data may be accessed for up to 10 years following the end of the study.
Access Criteria: Those who request the anonymous IPD must provide a plan of study explaining how the data will be used. Requests may be sent to the Central Contact Person. Requests will be reviewed based on the potential for the planned use of the IPD for advancing scientific knowledge and theory.

REFERENCES:
- [Derived] Mau T, Amin MR, Belafsky PC, Best SR, Friedman AD, Klein AM, Lott DG, Paniello RC, Pransky SM, Saba NF, Howard T, Dallas M, Patel A, Morrow MP, Skolnik JM. Interim Results of a Phase 1/2 Open-Label Study of INO-3107 for HPV-6 and/or HPV-11-Associated Recurrent Respiratory Papillomatosis. Laryngoscope. 2023 Nov;133(11):3087-3093. doi: 10.1002/lary.30749. Epub 2023 May 19. PMID 37204106

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT04398433/Prot_SAP_000.pdf